CLINICAL TRIAL: NCT00211822
Title: fMRI Studies in Pathological Gambling and Obsessive-Compulsive Disorder
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Studies in Pathological Gambling (PG) and Obsessive-Compulsive Disorder (OCD)
Status: Terminated | Type: Observational
Why Stopped: Enrollments closed after former PI Eric Hollander left institution. There are no results.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Abbott (Industry)
Responsible Party: Jennifer Bartz, PhD, Mount Sinai School of Medicine
Other Study IDs: GCO#04-1034
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Pathological Gambling; Obsessive Compulsive Disorder
Keywords: Pathological Gambling; Obsessive-Compulsive Disorder; Go No-go; Monetary incentives delay; fMRI
MeSH Terms: conditions — Gambling; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pathologic Gamblers
  Interventions: Procedure: fMRI
- Obsessive Compulsive Disorder
  Interventions: Procedure: fMRI
- Healthy Controls
  Interventions: Procedure: fMRI

INTERVENTIONS:
Procedure: fMRI — fMRI

SUMMARY:
This study will explore the brain processes associated with inhibition and reward processing in pathological gamblers and people with obsessive compulsive disorder compared to healthy controls.

DETAILED DESCRIPTION:
This study will explore the brain processes associated with inhibition and reward processing in pathological gamblers and people with obsessive compulsive disorder compared to healthy controls. Healthy participants and participants who are diagnosed with PG or OCD will undergo one fMRI scan. The brain scan will last about one and a half hours and will involve performing tasks while in the scanner.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults diagnosed with pathological gambling or obsessive compulsive disorder aged 18-55.
* Subject has signed an informed consent form
* Must provide contact information
* Must be in generally good health
* Must be willing and able to read written instructions and complete scales
* Must be English speaking
* In the opinion of the investigator, the subject is capable of complying with all study procedures

Pathological Gamblers only:

* Current diagnosis of pathological gambling, supported by DSM-IV SCI-PG
* Must score ≥ 5 on SOGS
* Must score ≥ 2 on item number 1 on the G-SAS
* Subjects must have a severity score of ≥ 4 (moderately ill) on the Clinical Global Impressions Scale - Severity (CGI-S)
* Must score ≥ 10 on questions 1-5 on PG-Y-BOCS
* Must score ≤ 15 on YMRS
* Must have gambled once within past 2 weeks of Screening Visit.

Exclusion Criteria:

* Subjects with a primary diagnosis of schizophrenia, personality disorder, or other psychotic disorders
* Subjects with a primary diagnosis of an Axis I disorder that may require intervention
* Must not score >24 on the Montgomery-Asberg Depression Rating Scale (MADRS) (pathological gamblers only)
* Subjects who live in a restrictive environment
* Subjects with a current DSM-IV diagnosis of substance dependence or abuse, excluding nicotine
* Subjects reporting a history of drug and/or alcohol dependence or abuse; subjects who report occasional drug use in the past will be discussed by a panel (consisting of Dr. Gilbert, Dr. Fan and Dr. Bartz), and will be considered for participation on a case by case basis
* Subjects who have used psychotropic medications in the past week to six weeks (depending on the medication)
* Subject has a positive drug urine screen
* Female subjects who are pregnant
* Subjects who report a history of severe liver, heart, or kidney disease because these conditions are associated with neurological sequella
* Employees of the investigator or study center or their families
* Finally, subjects who do not satisfy the following criteria will be excluded because they will be unable to undergo the MRI procedure. Specifically, subjects will be excluded who have:

  1. a pacemaker
  2. any implanted metallic chips in their head
  3. ever worked around a metal lathe or had a shrapnel (war or gun shot) wound/injury
  4. an implanted neuro-stimulatory or infusion/insulin pump
  5. any devices placed in their blood vessels
  6. any metal in/on their body
  7. kidney disease
  8. sickle-cell or hemolytic anemia
  9. claustrophobia
  10. any metallic tattoos
  11. any body piercing that cannot be removed
  12. dental braces
  13. any permanent make-up
  14. any cardiac stints

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2004-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
fMRI - go-nogo task | at baseline
  a measure of behavioral response inhibition
fMRI - monetary incentive delay (MID) task | at baseline
  a measure of neural response to anticipating and receiving monetary rewards

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States